CLINICAL TRIAL: NCT06470737
Title: Investigation of the Neurophysiological and Psychological Aspects of Itch
Brief Title: Investigation of Corticospinal Excitability Aspects of Itch and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20240004 1st subproject
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Itch; Pain
MeSH Terms: conditions — Pruritus; Pain | interventions — Saline Solution, Hypertonic; Histamine; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: we apply one of three experimental methods in your hand: either an injection of salt water (7% NaCl) or we apply small needles from the plant mucuna pruriens or histamine (1%) Histamine is an itch-provoking substance formed in the human body. For 10 minutes after this, you are to assess the itch and pain you perceive on a scale from 0 to 10, in which 0 is no itch/pain and 10 is worst itch/pain imaginable. We will also apply non-invasive magnetic stimulations to your brain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Other: Hypertonic Saline; Other: Histamine; Other: Cowhage; Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Other: Hypertonic Saline — A bolus injection of hypertonic saline (7% NaCl) will be administered to the FDI muscle using a 1 mL syringe with a disposable needle (27G), and the volume of the bolus will be 0.2 mL
Other: Histamine — A small drop of histamine dihydrochloride will be applied to a previously determined area on the volar forearm, followed by a prick through the drop
Other: Cowhage — This insertion is conducted by forceps using a stereo-microscope, and 30-35 spicules are gently rubbed into a 1 cm diameter skin area.
Device: Transcranial magnetic stimulation (TMS) — Transcranial magnetic stimulation (TMS) will be used to evoke motor-evoked potentials (MEPs) in the muscle of interest and cortical responses (TMS-evoked potentials - TEPs) in the motor cortex with a figure-eight-shaped cone coil.

SUMMARY:
The experiment consists of three experimental sessions conducted over a period of two weeks. In the first experimental session, we apply in your hand: either an injection of salt water (7% NaCl) or we apply small needles from the plant mucuna pruriens or histamine (1%). For 10 minutes after this, you are to assess the itch and pain you perceive. We will also apply non-invasive magnetic stimulations to your brain. During the experiment, you should fill in questionnaires. The second and third experimental sessions are conducted in the same way as the first session.

The purpose of this experiment is to investigate the changes appearing in the brain during artificially applied itch and pain corticomotor adaptations.

DETAILED DESCRIPTION:
The experiment consists of three experimental sessions conducted over a period of two weeks. The duration of each session is approx. two hours. In the first experimental session, we apply one of three experimental methods in your hand: either an injection of salt water (7% NaCl) or we apply small needles from the plant mucuna pruriens or histamine (1%) Histamine is an itch-provoking substance formed in the human body. For 10 minutes after this, you are to assess the itch and pain you perceive on a scale from 0 to 10, in which 0 is no itch/pain and 10 is worst itch/pain imaginable. We will also apply non-invasive magnetic stimulations to your brain. This is done using a magnetic coil which is held over your head. During the experiment, you should fill in questionnaires about how you experience itch/pain and about your personality. The second and third experimental sessions are conducted in the same way as the first session. However, we will apply one of the other two experimental methods than the one used in the first session (i.e., first session: histamine, second session: plant needles, third session: injection with salt water). The experimental methods will be applied in random order.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis), musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder (e.g., heart stroke), or psychiatric diagnoses (e.g. depression) that may affect the results
* Current use of medications that may affect the trial, such as antihistamines, antipsychotics, and painkillers, as well as systemic or topical steroids
* Skin diseases (e.g., atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Unable to pass the "Transcranial Magnetic Stimulation Adult Safety Screen" (subproject 1 and 2)
* Contraindications to transcranial magnetic stimulation (TMS) application (history of epilepsy, metal implants in head or jaw, etc.) (subproject 1 and 2)
* Presence of implanted hearing aids or metal implants on the face, including permanent makeup or tattoos (subproject 1 and 2)
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Numeric rating scales (NRS) | 1 minute after every itch/pain induction
  NRS are essentially VAS but have tick marks spaced every centimeter so as to create 11-point scale (from 0 to 10). Subject can use these tick marks as a guide when they mark their severity on the scale.
Measuring corticospinal excitability | Baseline
  Transcranial magnetic stimulation (TMS) will be used to evoke motor-evoked potentials (MEPs) in the muscle of interest and cortical responses (TMS-evoked potentials - TEPs) in the motor cortex with a figure-eight-shaped cone coil.
Measuring corticospinal excitability | 1 minute after every itch/pain induction for 10 minutes
  Transcranial magnetic stimulation (TMS) will be used to evoke motor-evoked potentials (MEPs) in the muscle of interest and cortical responses (TMS-evoked potentials - TEPs) in the motor cortex with a figure-eight-shaped cone coil.
Measuring corticospinal excitability | post induction (1 minute)
  Transcranial magnetic stimulation (TMS) will be used to evoke motor-evoked potentials (MEPs) in the muscle of interest and cortical responses (TMS-evoked potentials - TEPs) in the motor cortex with a figure-eight-shaped cone coil.
Measuring corticospinal excitability | post induction (30 minutes)
  Transcranial magnetic stimulation (TMS) will be used to evoke motor-evoked potentials (MEPs) in the muscle of interest and cortical responses (TMS-evoked potentials - TEPs) in the motor cortex with a figure-eight-shaped cone coil.
electromyography (EMG) recordings | 1 minute after every itch/pain induction
  For electromyography (EMG) recordings, two electrodes (Disposable Electrode Pack - AMBU Neuroline 720) will be placed on the muscle belly of the FDI muscle. The reference electrode will be placed on the ulnar styloid process of the left arm.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS). | Baseline
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale.
Itch Catastrophizing Scale (ICS). | Baseline
  he ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale.
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | Baseline
  The RST-PQ contains the following subscales: the Fight-Flight-Freeze System (FFFS, 10 items), which represents a defensive factor related to active avoidance of adverse stimuli; the Behavioral Inhibition System (BIS, 23 items), which represents a defensive factor related to anxiety and passive avoidance of adverse stimuli; and the Behavioral Approach System (BAS, 32 items), which reflects reward interest, goal-drive persistence, reward reactivity, and impulsivity. In total, 65 items have to be answered on a 4-point Likert-type scale
The Pittsburg Sleep Quality Index (PSQI) | Baseline
  The PSQI consists of 19 items generating seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The seven component scores can be summarized in a global score ranging from zero to 21 with higher scores reflecting a worse overall quality of sleep
Depression, Anxiety, Stress Scale (DASS-21) | Baseline
  he questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much".
Learned Helplessness Scale (LHS) | Baseline
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Positive And Negative Affect Schedule (PANAS) | Baseline
  PANAS measures positive and negative affect dimensions. Twenty words are associated with the subject's current feelings and have to be rated on a 5-points Likert-type scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No